CLINICAL TRIAL: NCT06936631
Title: REPLACE: the Impact of Catheter Replacement in Patients With Catheter-associated Urinary Tract Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, ecschippers, Coordinating investigator/ project leader, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL88486.058.25
Record Dates: First submitted 2025-03-24; First posted 2025-04-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Catheter Associated Urinary Tract Infection
Keywords: Catheter associated urinary tract infection; CAUTI; Urinary tract infection; UTI; Indwelling catheter; Urosepsis
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter replacement (Other): The control group undergoes catheter replacement within 3 days of starting antibiotic therapy. Choice of antibiotic agent follows standard care guidelines, with adjustments based on culture results.
  Interventions: Procedure: Catheter replacement
- Catheter retainment (Experimental): In the intervention group, the catheter is not replaced during CAUTI treatment. Choice of antibiotic agent follows standard careguidelines, with adjustments based on culture results. In this group, catheter replacement occurs according to the patient's regular schedule.
  Interventions: Procedure: Catheter retainment

INTERVENTIONS:
Procedure: Catheter replacement — In the intervention group, the catheter is not replaced during CAUTI treatment. Choice of antibiotic agent follows standard care guidelines, with adjustments based on culture results. In this group, catheter replacement occurs according to the patient's regular schedule.
  The control group undergoes catheter replacement within 3 days of starting antibiotic therapy. Choice of antibiotic agent follows standard care guidelines, with adjustments based on culture results.
  Arms: Catheter replacement
Procedure: Catheter retainment — In the intervention group, the catheter is not replaced during CAUTI treatment. Choice of antibiotic agent follows standard care guidelines, with adjustments based on culture results. In this group, catheter replacement occurs according to the patient's regular schedule. The control group undergoes catheter replacement within 3 days of starting antibiotic therapy. Choice of antibiotic agent follows standard care guidelines, with adjustments based on culture results.
  Arms: Catheter retainment

SUMMARY:
With this project the investigators aim to address the following question: "Is it beneficial to change bladder catheters during urinary tract infections?" There is debate regarding the usefulness of changing an indwelling catheter during antibiotic treatment of a catheter-associated urinary tract infection (CAUTI). The current guideline recommends catheter replacement, but is based on limited evidence. Our hypothesis is that there is no added value for patients to change the catheter during an antibiotic treatment for CAUTI. If refraining from catheter replacement is non inferior, this would result in a reduction of invasive procedures and reduction of healthcare associated costs. Patients with CAUTI and an indication for antibiotic treatment will be randomized to catheter replacement or no catheter replacement. The study will be conducted in academic and non-academic hospitals in The Netherlands. 300 patients will need to be included.

DETAILED DESCRIPTION:
As a result of the widespread application of urinary catheterization, catheter-associated urinary tract infection (CAUTI) is the most common healthcare associated infection. To fasten recovery and reduce the risk of a recurrent CAUTI, current guidelines recommend to replace the catheter at the onset of a CAUTI when the indwelling catheter has been in place for more than 2 weeks. This recommendation, however, is based on limited evidence. Additionally, there is significant practice variation in the Netherlands regarding catheter replacement in CAUTI. Given the limited evidence and significant practice variation in the Netherlands, this Randomized Controlled Trial including 300 CAUTI patients is needed.

The main question this study aims to answer is whether not changing the urinary catheter (catheter retainment) during a catheter-associated urinary tract infection (CAUTI) is non-inferior to catheter replacement in terms of the risk of a recurrent CAUTI within 90 days. Secondary objectives include 30-day mortality, health-related quality of life, time to resolution of CAUTI symptoms, complications of catheter replacement (e.g., discomfort, bleeding, sepsis) and healthcare and societal costs.

In the intervention group there will be no catheter replacement during CAUTI, meaning there will be no catheter replacement during the entire course of antibiotic treatment. In this group, catheter replacement will follow the patients regular replacement schedule, consequently meaning that it occurs outside the duration of the antibiotic treatment . The duration of antibiotic treatment is 10 days for both men and women. The control group follows the current guidelines. In this group, the catheter will be replaced within 3 days after the start of antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. An indwelling catheter, either a transurethral or suprapubic catheter, that has been in place for at least 2 weeks.
3. At least one CAUTI-related symptom, defined according to the IDSA guideline (11): onset or worsening of fever (> 38 degrees), rigors, altered mental status, malaise or lethargy with no other identified cause, flank pain, costovertebral angle tenderness, acute haematuria, pelvic discomfort, or suprapubic pain/tenderness. In patients with spinal cord injury, increased spasticity, autonomic dysreflexia, or sense of unease are also compatible with CAUTI.
4. Urine culture with ≥ 103 colony-forming units (CFU)/mL of ≥ 1 bacterial species, or urine culture with <103 CFU/mL along with a positive blood culture with the same microorganism as the urine culture.
5. The ability to provide written informed consent for the use of their data.
6. Sufficient proficiency in the Dutch or English language, both spoken and written, to effectively communicate with the research team and accurately complete the questionnaires.

Exclusion Criteria:

1. Having an immunodeficiency: High-dose corticosteroid use (any equivalent of ≥ 20 mg prednisolone per day for > 4 weeks), severe primary immunodeficiency, organ transplant, neutropenia (absolute neutrophil count < 0.50 x 10⁹/L)
2. Expiration of the indication of the indwelling catheter.
3. Having a planned (routine) catheter replacement during antibiotic therapy.
4. Contraindications for catheter replacement (judgement treating physician)
5. Kidney catheters (nephrostomy or double-J catheter).
6. Needing bladder irrigations because of gross haematuria.
7. Having bladder stones.
8. Female patients who are pregnant.
9. Having a life expectancy of < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Recurrent CAUTI within 90 days post-antibiotic treatment (T0 is the start of antibiotic treatment) | 90 days
  The definition of a recurrent CAUTI is identical to the definition used for inclusion. The pathogen does not have to be identical to the causative pathogen that was identified during the first episode. In case of a suspected recurrence, the following data will be collected: signs and symptoms, GCS, qSOFA, laboratory results, admission, antimicrobial treatment and treatment duration.

SECONDARY OUTCOMES:
Mortality | 180 days
  One of the secondary outcomes is 30-day mortality. However, if a patient passes away during the entire course of the study (180 days), this will be recorded.
Health-related quality of life measured using the PROMIS questionnaires | 90 days
  Health-related quality of life will be measured using the Patient-Reported Outcomes Measurement Information System Scale (PROMIS). This will measure various aspects of physical, mental, and social health. The PROMIS questionnaire will be administered at different times from baseline, to 90 days: baseline, day 3, day 7, day 28 and day 90.
Health-related quality of life measured using the EQ-5D-5L questionnaire | 180 days
  Health-related quality of life will be measured using the EQ-5D-5L questionnaire which assesses five dimensions of health-related quality of life: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The questionnaire will be administered at different times, from baseline, to 180 days: baseline, day 3, day 7, day 14, day 28, day 90 and day 180.
Time to resolution of CAUTI symptoms | 90 days
  After inclusion, patients are provided with a diary, in which they record their (CAUTI) symptoms. Additionally, the CAUTI-related symptoms are monitored by telephone at 3 days and then weekly from the start of antibiotic treatment until complete resolution of symptoms. Monthly telephone visits will also be conducted for optimal monitoring of recurrences, until the primary endpoint of 90 days.
Complications of catheter replacement | 3 days
  Complications of either catheter replacement or retainment and the severity of the complications will be recorded from the moment the procedure has taken place. A few examples of complications are discomfort, bleeding or sepsis. Considering the 3-day timespan between antibiotic initiation and catheter replacement, complications will be administered at 3 days.
Healthcare costs using a selection of items relevant for this population of the medical consumption (iMCQ) questionnaire | 90 days and 180 days
  Healthcare costs consist of the costs of the catheter replacement and other healthcare use of the patients. Cost of catheter replacement will be assessed using the micro costing approach in hospital setting. Other healthcare use (e.g. hospital days, cost of medication, outpatient visits, general practitioners visits, homecare visits) will be based on the iMCQ questionnaire administered to patients after 12 weeks and 6 months consisting of a selection of items relevant for this population.
Societal costs using a selection of items relevant for this population of the productivity (iPCQ) questionnaire | 90 days and 180 days
  Societal costs consisting of productivity losses in paid and unpaid work will be assessed using the iPCQ questionnaire administered to patients after 12 weeks and 6 months consisting of a selection of items of the relevant for this population.
Length of hospital stay and ICU-admission during hospital stay | 90 days
  If the patient presented at the hospital, it will be recorded whether admission occurred, and if so, whether the patient was admitted to a general ward or the intensive care unit. Additionally, if the patient is initially admitted to a general ward and subsequently transferred to the intensive care unit, this transfer will also be documented. The duration of the patient's admission will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, the data sharing plan will be developed.